CLINICAL TRIAL: NCT05314881
Title: Polymorphisms of the Tumor Necrosis Factor Superfamily 4 and Neutrophil Cytosolic Factor Gene in SLE Egyptian Patients.
Brief Title: NCF Gene & TNFSF4 in SLE Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmine Saad Makarem, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: gene polymorphism in SLE
Record Dates: First submitted 2022-03-26; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: System; Lupus Erythematosus
Keywords: TNFS4, NCF gene
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLE patients (Experimental)
  Interventions: Genetic: TNFS4, NCF gene

INTERVENTIONS:
Genetic: TNFS4, NCF gene — study the gene polymorphisms from the blood sample of the included SLE patients

SUMMARY:
the investigators objective is to identify the association of SNP polymorphisms in the TNFS4, and NCF gene and SLE Egyptian patients.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by clinical heterogeneity with variable severity. Among the SLE patients, two may share the same clinical manifestations but have different phenotypes.

This is why studies are searching for the different genes that might be associated with SLE susceptibility.

The Neutrophil cytosolic factor (NCF) Gene provide the instruction for the synthesis of group of proteins that form the NADPH oxidase enzyme complex, that is critical for the induction of reactive oxygen species (ROS) which in turn is important in the regulation of immune system.

While the Tumor necrosis factor superfamily 4 (TNFSF4) encodes the ligand for OX40 (OX40L), which delivers a strong costimulatory signal to activated effector T-cells and enhances both Th1 and Th2 responses when engaged with its receptor. Therefore, increased levels of cell surface OX40L may augment B cell differentiation and proliferation. The consequence of which is that the resulting autoantibodies and immune complexes cause disease pathology in SLE.

So, NCF and TNFSF4 gene polymorphism are supposed to be associated with SLE risk and pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients
* patients older than 18 years old

Exclusion Criteria:

* patients with other connective tissue diseases
* patients older than 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Concentration of gene polymorphism of the TNFS4 & NCF in SLE Egyptian patients. | 3 months
  Identify the number of Participants with SNP polymorphisms in the TNFS4, and NCF gene in SLE Egyptian patients and the relation between the concentration of polymorphism and disease activity

REFERENCES:
- [Background] Aziz MM, Galal MAA, Elzohri MH, El-Nouby F, Leong KP. Cross-cultural adaptation and validation of Systemic Lupus Erythematosus Quality of Life questionnaire into Arabic. Lupus. 2018 Apr;27(5):780-787. doi: 10.1177/0961203317747714. Epub 2018 Jan 7. PMID 29308728
- [Background] Kaiser R, Criswell LA. Genetics research in systemic lupus erythematosus for clinicians: methodology, progress, and controversies. Curr Opin Rheumatol. 2010 Mar;22(2):119-25. doi: 10.1097/BOR.0b013e3283361943. PMID 20035223
- [Background] Holmdahl R, Sareila O, Olsson LM, Backdahl L, Wing K. Ncf1 polymorphism reveals oxidative regulation of autoimmune chronic inflammation. Immunol Rev. 2016 Jan;269(1):228-47. doi: 10.1111/imr.12378. PMID 26683156
- [Background] Lu MM, Xu WD, Yang J, Ye QL, Feng CC, Li J, Pan HF, Tao JH, Wang J, Ye DQ. Association of TNFSF4 polymorphisms with systemic lupus erythematosus: a meta-analysis. Mod Rheumatol. 2013 Jul;23(4):686-93. doi: 10.1007/s10165-012-0708-8. Epub 2012 Aug 1. PMID 22850862
- [Background] Lane P. Role of OX40 signals in coordinating CD4 T cell selection, migration, and cytokine differentiation in T helper (Th)1 and Th2 cells. J Exp Med. 2000 Jan 17;191(2):201-6. doi: 10.1084/jem.191.2.201. No abstract available. PMID 10637265
- [Background] Ito T, Wang YH, Duramad O, Hanabuchi S, Perng OA, Gilliet M, Qin FX, Liu YJ. OX40 ligand shuts down IL-10-producing regulatory T cells. Proc Natl Acad Sci U S A. 2006 Aug 29;103(35):13138-43. doi: 10.1073/pnas.0603107103. Epub 2006 Aug 21. PMID 16924108
- [Background] Croft M. The role of TNF superfamily members in T-cell function and diseases. Nat Rev Immunol. 2009 Apr;9(4):271-85. doi: 10.1038/nri2526. PMID 19319144
- [Background] Stuber E, Neurath M, Calderhead D, Fell HP, Strober W. Cross-linking of OX40 ligand, a member of the TNF/NGF cytokine family, induces proliferation and differentiation in murine splenic B cells. Immunity. 1995 May;2(5):507-21. doi: 10.1016/1074-7613(95)90031-4. PMID 7749983
- [Background] Olsson LM, Johansson AC, Gullstrand B, Jonsen A, Saevarsdottir S, Ronnblom L, Leonard D, Wettero J, Sjowall C, Svenungsson E, Gunnarsson I, Bengtsson AA, Holmdahl R. A single nucleotide polymorphism in the NCF1 gene leading to reduced oxidative burst is associated with systemic lupus erythematosus. Ann Rheum Dis. 2017 Sep;76(9):1607-1613. doi: 10.1136/annrheumdis-2017-211287. Epub 2017 Jun 12. PMID 28606963